CLINICAL TRIAL: NCT05549921
Title: TAEST16001 in Patients With Soft Tissue Sarcoma With Positive NY-ESO-1 Expression (Genotype: HLA-A*02:01): an Multi-center, Open-label and Single Arm Phase II Study
Brief Title: Phase II Study of TAEST16001 in Soft Tissue Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Guangdong Xiangxue Precision Medical Technology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xing Zhang, Director of department of sarcoma and melanoma, Principal Investigator, Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAEST16001 Phase II
Record Dates: First submitted 2022-09-04; First posted 2022-09-22 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NY-ESO-1 TCR Specific T cell Therapy (Experimental): This research is divided into two stages, Stage 1 and Stage 2, respectively. In Stage 1, 14 patients with advanced soft tissue sarcoma with positive expression of tumor antigen NY-ESO-1 and HLA-A*02:01 genotype were enrolled. A further 42 patients will be enrolled in Stage 2, where the primary efficacy analysis will be performed at 3 months after the completion of cell reinfusion in the last subject, with a target ORR of 25%.
  Interventions: Biological: NY-ESO-1(TCR Affinity Enhancing Specific T cell Therapy)

INTERVENTIONS:
Biological: NY-ESO-1(TCR Affinity Enhancing Specific T cell Therapy) — NY-ESO-1(TCR Affinity Enhancing Specific T cell Therapy)

SUMMARY:
The main purpose of this trial is to evaluate the efficacy and safety of TAEST16001 cells in the treatment of advanced soft tissue sarcoma patients with HLA-A*02:01 tissue genotype and positive tumor antigen NY-ESO-1 expression.

DETAILED DESCRIPTION:
This is a single-arm, open label, multi-center, phase II study. The investigators include advanced soft tissue sarcoma with failure in standard treatment or no recommended standard therapy.

TCR-T cell therapy has made a breakthrough for tumors in recent years. Phase I/II trial of NY-ESO-1-specific TCR-T treatment for synovial sarcoma and melanoma, conducted by the Rosenberg team at the National Cancer Institute, showed that 61% Synovial cell sarcoma patients and 55% melanoma patients benefit from this treatment, without severe side effects found in T cell receptor (TCR) transduced T-Cell Immunotherapy.

This clinical trial is mainly focused on cancer-testis antigen, because it is not expressed in normal cells. NY-ESO-1 antigen as one member of cancer-testis antigen, is commonly expressed in 10-50% of melanoma, lung, liver, esophageal, breast, prostate, bladder, thyroid and ovarian cancer cases, 60% of multiple myeloma cases, and 70-80% of synovial sarcoma. NY-ESO-1 expression was also found in 88.2% of myxoid liposarcomas, 61.1% of synovial sarcomas, 31.3% of osteosarcomas, 21.4% of pleomorphic liposarcomas, 16.7% of desmoplastic small round cell tumors, and 14.3% of chondrosarcomas. Although the NY-ESO-1 TCR cell therapy for synovial sarcoma and melanoma has benefited many patients and the phase I trial has been performed, its effect and safety on advanced soft tissue sarcoma is still unknown.

The patients must meet the two criteria: HLA-A*0201positive and NY-ESO-1 positive cells≥20% by immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* Before any research-related operations, they should sign the informed consent Consent Form (ICF) (Genotype and Tumor Antigen Screening and Primary Screening);
* Age ≥18 years, and ≤70 years;
* His/cytology confirmed, unresectable or metastatic soft tissue sarcoma;
* The current stage is the failure of standard treatment (disease progression or recurrence or intolerance, such as chemotherapy, radiotherapy, targeted therapy, etc.) or lack of effective treatment methods, specifically: In addition to acinar soft tissue sarcoma and for pathological subtypes other than epithelioid sarcoma, at least adriamycin or doxorubicin combined with ifosfamide standard chemotherapy regimen should fail or not tolerate chemotherapy; For acinar soft tissue sarcoma and epithelioid sarcoma, need failure or intolerance of previous targeted drugs [anti-angiogenesis such as Anlotinib, pazopanib, etc.]; Note: Treatment failure refers to disease progression or inability during treatment or within 3 months of the last treatment Tolerable; disease progression in patients with neoadjuvant or adjuvant therapy > 6 months after the end of treatment can be considered first-line therapy;
* At least 1 measurable lesion (according to RECIST1.1 criteria [see Appendix 4 for details]);
* Genotype and tumor antigen screening must meet the following 2 criteria: HLA-A*02:01 positive; NY-ESO-1* positive: immunohistochemical staining positive cells are ≥20%;
* ECOG score of 0-1 and expected survival period of more than 3 months;
* Echocardiography showed left ventricular ejection fraction ≥ 50%;
* Laboratory test results should at least meet the following specified indicators: White blood cell count ≥ 3.0×109 /L; Absolute neutrophil count (ANC) ≥ 1.5×109/L (without G-CSF and GM-CSF support, at least 14 days before lymphadenectomy); Absolute lymphocyte count (ALC) ≥ 0.7× 109/L; Platelet (PLT) ≥ 75×109/L (no blood transfusion therapy 14 days before lymphadenectomy chemotherapy); hemoglobin ≥ 9 g/dL (no blood transfusion therapy 14 days before lymphoid clearing chemotherapy); Coagulation International Normalized Ratio (INR) ≤ 1.5×ULN unless anticoagulant therapy;Partial prothrombin time (APTT) ≤ 1.5×ULN unless anticoagulant therapy; Serum creatinine ≤ 1.5 mg /dL (or 132.6 μmol/L); Creatinine clearance ≥60 mL/min; Aspartate aminotransferase (AST/SGOT)≤2.5×ULN; Alanine aminotransferase (ALT/SGPT)≤2.5×ULN; Total bile red Prime (TBIL)≤1.5×U LN; Note: If patients with liver metastases or patients with primary liver tumor lesions, aspartate aminotransferase and alanine aminotransferase should be ≤5× ULN;
* Females of childbearing age who have not received sterilization before menopause must agree to be removed from the study treatment (clearing). effective contraceptive measures should be used from the beginning of the last cell infusion to one year after the last cell infusion, and the serum pregnancy test was negative within 14 days before the first cell infusion; ) and up to one year after the last cell infusion, use effective contraception.

Exclusion Criteria:

* Received the last leukocyte apheresis within 4 weeks. Anti-tumor therapy (chemotherapy, endocrine therapy, targeted therapy, tumor embolization or traditional Chinese medicine with anti-tumor indications, etc.); immunotherapy within 1 month before the signing of the main informed consent;
* 4 days before cell infusion received live attenuated vaccine within 1 week;
* Patients with ≥3 bone metastases;
* Known to have allergic reactions to any components used in the treatment of this study;
* No previous surgery or treatment-related adverse reactions recovered to <Grade 2 CTCAE v5.0;
* Patients with a history of meningeal metastasis or central nervous system metastasis, or patients with clear underlying diseases of the central nervous system within 6 months before cell reinfusion, and left significant symptoms;
* Uncontrolled hypertension (systolic blood pressure >160 mmHg and/or diastolic blood pressure >90 mmHg) or clinically significant (eg active) cardiovascular and cerebrovascular diseases, such as cerebrovascular accident within 1 month), myocardial infarction (within 6 months before signing the main informed consent), unstable angina, congestive heart failure with New York Heart Association (NYHA) class II or above, or severe arrhythmia that cannot be treated with drugs Control or have potential impact on study treatment; ECG results show clinically significant abnormality or average QTcF ≥ 450 ms in 3 consecutive times (at least 5 minutes between each time) (see Appendix 2 for the formula);
* Combined with other serious devices;
* Patients with systemic active infections that require treatment, including but not limited to active tuberculosis, known HIV-positive patients or clinically active hepatitis A, B, and C patients, including virus carriers;
* Patients with autoimmune diseases: those with a history of inflammatory bowel disease and a history of autoimmune diseases judged by the investigator to be unsuitable for this study, such as systemic lupus erythematosus, vasculitis, and infiltrative lung disease, should be excluded ( (except for vitiligo and psoriasis that do not require systemic immunosuppressive therapy);
* G-CSF or GM-CSF has been used within 2 weeks before leukapheresis, or within 4 weeks before cell reinfusion and planned to be used during the study period (If there is long-term use) systemic cortisone steroids, hydroxyurea, immunomodulatory drugs (eg: alpha or gamma interferon, GM-CSF, mTOR inhibitors, cyclosporine, thymosin, etc.);
* Organ isotypes History of transplantation, allogeneic stem cell transplantation and renal replacement therapy;
* Known uncontrolled diabetes, pulmonary fibrosis, interstitial lung disease, acute lung disease or liver failure;
* Known alcohol and/or drug abuser;
* Pregnant or lactating women;
* Suffering from any co-existing medical conditions or diseases that the investigators determined may affect the conduct of this trial.
* Subjects with no legal capacity/restricted capacity;
* Previously received treatment targeting NY-ESO-1, or received cellular immunotherapy within 12 months before cell reinfusion, investigator Patients deemed unsuitable for enrollment;
* Received immunotherapy (immune checkpoint blockade therapy: such as PD-1, PD-L1 antibody treatment, etc.) within 3 months before cell reinfusion;
* Patients judged by the investigator Difficulty completing all visits or procedures (including follow-up periods) required by the study protocol, or insufficient compliance to participate in this study; or patients deemed unsuitable for inclusion by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-07-08 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 270 days
  The objective response rate (ORR), as assessed by an independent imaging evaluation committee (IRC), was used as the endpoint (response evaluation criteria based on solid tumors, version 1.1 [RECIST1.1]) to evaluate the TAEST16001 cell therapy tissue genotype as HLA-A*02:01 and tumor antigen NY-ESO-1 Efficacy of positive expression in patients with advanced soft tissue sarcoma.

SECONDARY OUTCOMES:
Disease control rate (DCR) | 270 days
  Assessed by in all patients with advanced soft tissue sarcoma who received TAEST16001 cell reinfusion, according to RECIST.
Progression-free survival (PFS) | 270 days
  Assessed by in all patients with advanced soft tissue sarcoma who received TAEST16001 cell reinfusion.
Duration of response (DOR) | 270 days
  Assessed by in all patients with advanced soft tissue sarcoma who received TAEST16001 cell reinfusion, according to RECIST.
Time to tumor response (TTR) | 270 days
  Assessed by in all patients with advanced soft tissue sarcoma who received TAEST16001 cell reinfusion, according to RECIST.
Overall survival (OS) | 270 days
  Assessed by IRC and investigator in all patients with advanced soft tissue sarcoma who received TAEST16001 cell reinfusion.
Number of participants with other abnormal laboratory values and/or adverse events that are related to treatment | 270 days
  According to CTCAE 5.0 criteria.
Maximum Plasma Concentration (Cmax) | 270 days
  To observe the proliferation and persistence of TAEST16001 cells in vivo.
Maximum time to peak (Tmax) | 270 days
  To observe the proliferation and persistence of TAEST16001 cells in vivo.
Activity of T lymphocyte subsets | 270 days
  To observe the influence of TAEST16001 cells on human immunological activity.
Activity of peripheral blood antigen specific cytotoxic lymphocyte (CTL) | 270 days
  To observe the influence of TAEST16001 cells on human immunological activity.
Activity of effector T cells | 270 days
  To observe the influence of TAEST16001 cells on human immunological activity.
Life quality scale | 270 days
  According to European Organization for Research on Treatment of Cancer (EORTC) QLQ-C30 life quality scale, 30 items were divided into 5 functional domains (physical, role, cognitive, emotional and social functions), 3 symptom domains (fatigue, pain, nausea and vomiting), 1 general health/quality of life domain and 6 single domains. The score for each domain is obtained by summing the scores of items included in each domain and dividing by the number of items included. The final total scores range from 0 to 100 by standardizing the conversion of the raw scores. Higher scores in the functional and general health domains indicate better functioning and quality of life, and higher scores in the symptom domain indicate more symptoms or problems (worse quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Xing Zhang, PhD, MD, Principal Investigator — Sun Yat-sen University
Locations (2):
- China (2):
  - Sun Yat-Sen Univerisity Cancer Center, Guangzhou, Guangdong
  - Peking University Cancer Hospital & Institute, Beijing